CLINICAL TRIAL: NCT01763307
Title: A Phase II Randomized, Double Blind, Placebo Study to Evaluate the Efficacy of Vitamin K1 Cream Treatment Compared to Placebo for the Prevention of Papulo-pustular Rash in Metastatic Colorectal Patients Receiving First Line EGFRI Treatment.
Brief Title: A Study to Examine the Effect of Reconval K1 Cream to Prevent Skin Toxicity From EGFRI
Acronym: EGFRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EGFRI-MER-1a-HMO-CTIL
Record Dates: First submitted 2012-12-24; First posted 2013-01-08 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2017-08

CONDITIONS: Rash Due to Epidermal Growth Factor Receptor Inhibitors
Keywords: EGFRI; COLON CANCER; SKIN TOXICITY; RECONVAL K1 cream
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RECONVAL CREAM (Experimental): half face treated with RECONVAL CREAM
  Interventions: Drug: RECONVAL CREAM
- PLACEBO (Placebo Comparator): half face treated with PLACEBO cream
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: RECONVAL CREAM
  Arms: RECONVAL CREAM
Drug: PLACEBO
  Arms: PLACEBO

SUMMARY:
Vitamin K1 cream may prevent papulopustular rash induced by EGFRI given to metastatic colorectal cancer patients.

This study will prospectively accrue metastatic colorectal patients receiving EGFRI and treat with reconval cream half face versus placebo cream half face to study whether Vitamin k1 cream can prevent the typical skin eruption caused by EGFRI.

ELIGIBILITY:
Inclusion Criteria:

* metastatic colon cancer patients
* male or female
* age> 18
* treated EGFRI

Exclusion Criteria:

* prior treatment with EGFRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Potential reduction in skin toxicity by Vitamin K1 cream in metastatic colorectal patients treated with EGFRI | 12 weeks
  Reduction in numbers of papulo-pustular eruptions in the treatment fields compared to the placebo treated side. Changes in follicular eruptions, dryness/redness of skin estimated by the grading scale developed by the Multinational Association of Supportive Care in Cancer (MASCC) skin toxicity study group 4.0. Patients own experience of efficacy estimated by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Merims, MD, Principal Investigator — Hadassah Medcial Organization